CLINICAL TRIAL: NCT02791100
Title: Promotion of Egg and Eggshell Powder Consumption Improve Nutritional Status of Children of Under Two Years of Age: A Cluster Randomized Controlled Community Trial in Halaba Ethiopia
Brief Title: Promotion of Egg and Eggshell Powder Consumption Improve Nutritional Status of Children in Halaba Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Hawassa University (Other)
Responsible Party: Principal Investigator, Susan Whiting, Ph.D., University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HU-UoS-EGG
Record Dates: First submitted 2015-09-21; First posted 2016-06-06 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Thinness; Food Habits; Health Knowledge, Attitudes, Practices
Keywords: height; weight; diet; complementary foods; protein; calcium
MeSH Terms: conditions — Thinness; Feeding Behavior; Behavior; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No promotion of chicken eggs (No Intervention): The community receives no chickens and therefore has no additional eggs or egg shell powder for children
- Promotion of Chicken eggs for children (Experimental): The community receives chickens so that each study child receives 2 eggs a day and also receives some egg shell daily (1/4 bottle cap which provides 500 mg Ca). The community receives information on using the egg and eggshell, and has help in caring for the chickens.
  Interventions: Behavioral: Promotion of chicken eggs

INTERVENTIONS:
Behavioral: Promotion of chicken eggs — Community is provided with chickens and young children are to receive 2 eggs a day plus egg shell
  Arms: Promotion of Chicken eggs for children

SUMMARY:
Young children in Ethiopia lack sufficient protein and micronutrients for growth and development. The overall purpose is to assess the effects of promoting egg and eggshell powder consumption on improving the nutritional status of children 6 to 15 months in Halaba Special Woreda, Southern Ethiopia. The hypothesis is that providing chickens to produce eggs (egg and eggshell) for young children will improve growth in otherwise malnourished young children. Upon providing chickens, the nutritional status of young children prior and after the intervention (by 6 months) will be assessed. Identification of the knowledge, attitude and practices (KAP) of mothers on egg and eggshell powder consumption by their children before and after the intervention in the intervention group will be done. Caregivers will be instructed to give each child 1 egg (cooked) and 1/4 "bottle cap" of eggshell (500 mg calcium) per day in the intervention. Hemoglobin will be measured as an indicator of overall nutritional status. Throughout the study, any problems arising in keeping chickens will be recorded in order to assess the feasibility and practicality of raising chickens as way to improve nutritional status of young children. The study is novel in that investigators are providing a way to have increased protein, increased micronutrients, and use of eggshell as a source of calcium.

DETAILED DESCRIPTION:
Young children in Ethiopia lack sufficient protein and micronutrients for growth and development.The study will adopt a 6-month cluster-randomized and controlled trial design. There will be a treatment group (communities receiving chickens) and a control group (no chickens for the 6 months of the study).

Study participants will be recruited from all children aged between 6-15 months old, who are residents of 6 Kebeles in the clusters. from these 6, the Control and Intervention areas will be randomly selected. This age group is selected because it is the time of introduction of complementary food and it will be easier to see the clear effect of egg on the children growth, rather than choosing older children.

In the Intervention group, children who are known to be allergic to egg will be excluded from the study. The following measurements will be made at baseline (prior to chicken ceremony in intervention areas) and at month 6: dietary assessment by 24-hour recall of child and mother; food frequency questionnaire for diet diversity score; hemoglobin test (involving a single finger prick) of child; weight and height (or for very young children, length); knowledge and attitude questions on egg and egg-shell nutrition. At baseline only, caregivers will answer demographic questions. Monthly, there will be monitoring of egg and eggshell consumption by children as well as measurement of height (length), and a structured questionnaire on morbidity. In the intervention group, caregivers will be instructed to provide one egg and a small amount of eggshell (providing 500 mg calcium). At 9 month, the research assistant will visit the Intervention communities to informally gather data on chickens being used, participant children's health status (any follow-up morbidity data). Throughout data will be collected on infection rate, with the possibility of improvement due to better nutrition but also awareness that bringing chickens into the community could pose a risk to very young children. As well, there will be formal follow-up observation at one community site with focus group discussion and key informant interviews, as a way to assess feasibility and practically of chicken donation in the future. This will be a convenience sample representing participant parents, community leaders, Agriculture Extension workers, Health extension workers, persons who were not directly involved. Those targeted for interviews will be the extension workers from whom feedback will be provided, while focus groups will be held with others who are able to attend a focus group session .

Data checks will be provided by the MSc student and his local supervisor who planned the study but is not directly involved in day-to-day running of the intervention. The student will write SOPs for all procedures. Missing data will be accounted for but as this is a community based study group means will be used for most outcome measurements. Comparing of two means/the differences of means between the intervention and control groups will be done using independent two sample t-test. Continuous outcomes will be analyzed using paired t-test. Bivariate analysis will be used to see the overall effect of independent variables and then further multivariate analysis (multiple linear regressions) will be done to see the effect of each independent variable. Both crude and adjusted risk ratio with 95% confidence interval will be reported. Other variables and relevant findings will be also analyzed using proper statistical test/analysis techniques and reported accordingly. P-value of less than 0.05 will be taken as significant

ELIGIBILITY:
Inclusion Criteria:

* not known to be allergic to eggs.
* not undergoing therapy for moderate or severe malnutrition.

Exclusion Criteria:

* children undergoing treatment for malnutrition

Ages: 6 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
weight (kg) | 6 months
  weight (kg) of child

SECONDARY OUTCOMES:
knowledge, attitudes and practices on egg and egg shell use via questionnaire | 6 months
  Via questionnaire assess whether mothers have improved complementary feeding
health status as hemoglobin measure | 6 months
  measure hemoglobin as measure of overall health status
incidence of reported infections in study children | 6 months
  record number of reported infections

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Whiting, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Hawassa University School of Nutrition, Food Science, Awasa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Only group data, means, median

REFERENCES:
- [Background] Brun LR, Lupo M, Delorenzi DA, Di Loreto VE, Rigalli A. Chicken eggshell as suitable calcium source at home. Int J Food Sci Nutr. 2013 Sep;64(6):740-3. doi: 10.3109/09637486.2013.787399. Epub 2013 Apr 22. PMID 23607686
- [Background] Mukaratirwa S, Khumalo MP. Prevalence of helminth parasites in free-range chickens from selected rural communities in KwaZulu-Natal province of South Africa. J S Afr Vet Assoc. 2010 Jun;81(2):97-101. doi: 10.4102/jsava.v81i2.113. PMID 21247015
- [Background] Victora CG, de Onis M, Hallal PC, Blossner M, Shrimpton R. Worldwide timing of growth faltering: revisiting implications for interventions. Pediatrics. 2010 Mar;125(3):e473-80. doi: 10.1542/peds.2009-1519. Epub 2010 Feb 15. PMID 20156903
- [Background] Negash C, Belachew T, Henry CJ, Kebebu A, Abegaz K, Whiting SJ. Nutrition education and introduction of broad bean-based complementary food improves knowledge and dietary practices of caregivers and nutritional status of their young children in Hula, Ethiopia. Food Nutr Bull. 2014 Dec;35(4):480-6. doi: 10.1177/156482651403500409. PMID 25639132
- [Result] Omer A, Mulualem D, Classen H, Vatanparast H, Whiting SJ (2018) Promotion of Egg and Eggshell Powder Consumption Improves Nutritional Status of Children of Under Two Years of Age: A Cluster Randomized Controlled Community Trial in Halaba Sp. Woreda, SNNPR Journal of Agricultural Science, 10(5), ISSN 1916-9752 E-ISSN 1916-9760.